CLINICAL TRIAL: NCT05582226
Title: A Randomized, Single Blinded Study of the Augmentation of Anterior Cruciate Ligament Reconstruction Using Stump-Derived Mesenchymal Stem Cells Versus Standard of Care Anterior Cruciate Ligament Reconstruction
Brief Title: Augmentation of Anterior Cruciate Ligament Reconstruction Using Mesenchymal Stem Cells and Collagen Matrix Carrier
Acronym: BioACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioACL2.0
Record Dates: First submitted 2022-10-06; First posted 2022-10-17 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of two groups, the first group receiving stump stem cell infusion and the second group receiving standard of care ACL reconstruction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL reconstruction utilizing stump-derived mesenchymal stem cells (Experimental): This is the test group of this study. These participants will receive the augmented ACL reconstruction treatment involving extraction and injection of mesenchymal stem cells. Stem cell tissue will be harvested from each participant using the GraftNet device intraoperatively. During the intra-articular preparation phase of the reconstruction, the stem cell tissue will be applied to the ACL graft using a bovine collagen matrix.
  Interventions: Procedure: ACL reconstruction; Procedure: Mesenchymal stem cell implantation
- Standard of care ACL reconstructive surgery (Other): This is the control group of this study. These participants will receive standard ACL reconstructive surgery without any augmentations.
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — Orthopedic surgical operation in which a ruptured anterior cruciate ligament is repaired and reattached to the muscle connection points with a "graft", a fashioned ligament that is meant to serve as a replacement for the ruptured muscle tissue.
Procedure: Mesenchymal stem cell implantation — Stem cells are to be extracted from tissue at the stump of the ACL attachment point and inserted on the graft in the hopes of improving healing response
  Arms: ACL reconstruction utilizing stump-derived mesenchymal stem cells

SUMMARY:
The goal of this observational study is to compare patient outcomes for reconstructive surgery of ACL tears. This study utilizes two randomized groups, one being the control group that receives standard ACL reconstructive surgery, while the other is the test group at will receive an injection of stem cells taken from elsewhere within the body. The main objectives are to determine the usefulness of stem cells as a cost-effective implant in reconstructive surgery and to determine if the stem cells provide more optimized healing outcomes.

Participants will:

* Receive ACL reconstructive surgery as normal
* One-half of the participants will receive stem cells at the repair site as the test group
* All participants will have 3, 6, 9, 12, 18, and 24 month followups to chart their recovery progress Thus, the outcomes of the group receiving stem cell injections will be compared directly with the outcomes of the standard ACL reconstructive care group.

DETAILED DESCRIPTION:
The primary objective of this study is to develop a cost-effective, autologous biologic augmentation technique for ACL reconstruction. The technique involves encasing MSCs harvested from the patient's ACL stump tissue with the GraftNet device in a porous bovine collagen matrix carrier around the ACL autograft. This study is key to determining a reproducible and effective autologous biologic augmentation technique that can be utilized at the point-of-care during ACL reconstruction surgery.

FTA results as well as measurements from MRI evaluation will be recorded and utilized to quantify the healing and ACL graft maturation processes. MRI evaluation will be performed in accordance with accepted ACL imaging protocols. This data will then be compared to FTA results and MRI evaluation from patients who did not undergo the bioaugmentation technique for ACL reconstruction.

Study design will be a prospective, blinded randomized, single center trial. Patients at the Andrews Institute who meet the inclusion criteria will have the study explained in detail and informed consent will be obtained as outlined below. Fifty patients will be blinded, randomized, and undergo a Bone-Patellar Tendon-Bone (BTB) ACL reconstruction surgery. Twenty-Five randomized patients will receive standard of care (SOC) BTB ACL reconstruction surgery. Twenty-Five randomized patients will receive BTB ACL reconstruction surgery augmented with the patient's ACL stump tissue harvested with the GraftNet device and a porous bovine collagen matrix carrier around the ACL autograft.

At each follow up visit after ACL reconstruction, patient reported outcome measures (PROMs) will be collected by the research team to assist in assessing the overall health and rehabilitation of each participant. The following patient reported outcomes will be collected in written or electronic format after informed consent has been obtained from each participant:Tampa Scale of Kinesiophobia, International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC), Patient Reported Outcome Measurements Information System (PROMIS), Single Assessment Numeric Evaluation (SANE), and Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 14 and 50 who are scheduled to have ACL reconstruction by one of the investigating physicians

Exclusion Criteria:

* Patients requiring ACL and posterior cruciate ligament combined surgery
* Patients with a history of an autoimmune disease, diabetes, a blood/clotting disorder
* History of previous surgery on the injured knee
* Patients outside of the acceptable age range of this study

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-08-16 (Estimated); Study Completion 2023-08-16 (Estimated)

PRIMARY OUTCOMES:
Assessing functional movement using Functional Testing Algorithm | 3 months post-operative
  Battery of tests used to determine the participant's capability of movement during the post-op recovery process; provides physical functional evidence of biomechanical recovery
Assessing functional movement using Functional Testing Algorithm | 6 months post-operative
  Battery of tests used to determine the participant's capability of movement during the post-op recovery process; provides physical functional evidence of biomechanical recovery
Assessing functional movement using Functional Testing Algorithm | 9 months post-operative
  Battery of tests used to determine the participant's capability of movement during the post-op recovery process; provides physical functional evidence of biomechanical recovery
Assessing functional movement using Functional Testing Algorithm | 12 months post-operative
  Battery of tests used to determine the participant's capability of movement during the post-op recovery process; provides physical functional evidence of biomechanical recovery
Assessing functional movement using Functional Testing Algorithm | 18 months post-operative
  Battery of tests used to determine the participant's capability of movement during the post-op recovery process; provides physical functional evidence of biomechanical recovery
Assessing functional movement using Functional Testing Algorithm | 24 months post-operative
  Battery of tests used to determine the participant's capability of movement during the post-op recovery process; provides physical functional evidence of biomechanical recovery

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- Andrews Research and Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffin LY, Agel J, Albohm MJ, Arendt EA, Dick RW, Garrett WE, Garrick JG, Hewett TE, Huston L, Ireland ML, Johnson RJ, Kibler WB, Lephart S, Lewis JL, Lindenfeld TN, Mandelbaum BR, Marchak P, Teitz CC, Wojtys EM. Noncontact anterior cruciate ligament injuries: risk factors and prevention strategies. J Am Acad Orthop Surg. 2000 May-Jun;8(3):141-50. doi: 10.5435/00124635-200005000-00001. PMID 10874221
- [Background] Gianotti SM, Marshall SW, Hume PA, Bunt L. Incidence of anterior cruciate ligament injury and other knee ligament injuries: a national population-based study. J Sci Med Sport. 2009 Nov;12(6):622-7. doi: 10.1016/j.jsams.2008.07.005. Epub 2008 Oct 2. PMID 18835221
- [Background] Leathers MP, Merz A, Wong J, Scott T, Wang JC, Hame SL. Trends and Demographics in Anterior Cruciate Ligament Reconstruction in the United States. J Knee Surg. 2015 Oct;28(5):390-4. doi: 10.1055/s-0035-1544193. Epub 2015 Jan 30. PMID 25635874
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770
- [Background] Ullah I, Subbarao RB, Rho GJ. Human mesenchymal stem cells - current trends and future prospective. Biosci Rep. 2015 Apr 28;35(2):e00191. doi: 10.1042/BSR20150025. PMID 25797907
- [Background] Anz AW, Branch EA, Rodriguez J, Chillemi F, Bruce JR, Murphy MB, Suzuki RK, Andrews JR. Viable Stem Cells Are in the Injury Effusion Fluid and Arthroscopic Byproducts From Knee Cruciate Ligament Surgery: An In Vivo Analysis. Arthroscopy. 2017 Apr;33(4):790-797. doi: 10.1016/j.arthro.2016.09.036. Epub 2016 Dec 30. PMID 28043750
- [Background] Branch EA, Matuska AM, Plummer HA, Harrison RM, Anz AW. Platelet-Rich Plasma Devices Can Be Used to Isolate Stem Cells From Synovial Fluid at the Point of Care. Arthroscopy. 2021 Mar;37(3):893-900. doi: 10.1016/j.arthro.2020.09.035. Epub 2020 Oct 1. PMID 33010328
- [Background] Shi Y, Zhang X, Wan Z, Liu X, Chen F, Zhang J, Leng Y. Mesenchymal stem cells against intestinal ischemia-reperfusion injury: a systematic review and meta-analysis of preclinical studies. Stem Cell Res Ther. 2022 May 26;13(1):216. doi: 10.1186/s13287-022-02896-y. PMID 35619154
- [Background] Fu X, Liu G, Halim A, Ju Y, Luo Q, Song AG. Mesenchymal Stem Cell Migration and Tissue Repair. Cells. 2019 Jul 28;8(8):784. doi: 10.3390/cells8080784. PMID 31357692
- [Background] Kim MJ, Son MJ, Son MY, Seol B, Kim J, Park J, Kim JH, Kim YH, Park SA, Lee CH, Lee KS, Han YM, Chang JS, Cho YS. Generation of human induced pluripotent stem cells from osteoarthritis patient-derived synovial cells. Arthritis Rheum. 2011 Oct;63(10):3010-21. doi: 10.1002/art.30488. PMID 21953087
- [Background] Matsumoto T, Ingham SM, Mifune Y, Osawa A, Logar A, Usas A, Kuroda R, Kurosaka M, Fu FH, Huard J. Isolation and characterization of human anterior cruciate ligament-derived vascular stem cells. Stem Cells Dev. 2012 Apr 10;21(6):859-72. doi: 10.1089/scd.2010.0528. Epub 2011 Aug 17. PMID 21732814
- [Background] Mifune Y, Matsumoto T, Takayama K, Terada S, Sekiya N, Kuroda R, Kurosaka M, Fu FH, Huard J. Tendon graft revitalization using adult anterior cruciate ligament (ACL)-derived CD34+ cell sheets for ACL reconstruction. Biomaterials. 2013 Jul;34(22):5476-87. doi: 10.1016/j.biomaterials.2013.04.013. Epub 2013 Apr 28. PMID 23632324
- [Background] Suzuki S, Muneta T, Tsuji K, Ichinose S, Makino H, Umezawa A, Sekiya I. Properties and usefulness of aggregates of synovial mesenchymal stem cells as a source for cartilage regeneration. Arthritis Res Ther. 2012 Jun 7;14(3):R136. doi: 10.1186/ar3869. PMID 22676383
- [Background] Horie M, Driscoll MD, Sampson HW, Sekiya I, Caroom CT, Prockop DJ, Thomas DB. Implantation of allogenic synovial stem cells promotes meniscal regeneration in a rabbit meniscal defect model. J Bone Joint Surg Am. 2012 Apr 18;94(8):701-12. doi: 10.2106/JBJS.K.00176. PMID 22517386
- [Background] Koyama N, Okubo Y, Nakao K, Osawa K, Fujimura K, Bessho K. Pluripotency of mesenchymal cells derived from synovial fluid in patients with temporomandibular joint disorder. Life Sci. 2011 Nov 7;89(19-20):741-7. doi: 10.1016/j.lfs.2011.09.005. Epub 2011 Sep 19. PMID 21958469
- [Background] Harvanova D, Tothova T, Sarissky M, Amrichova J, Rosocha J. Isolation and characterization of synovial mesenchymal stem cells. Folia Biol (Praha). 2011;57(3):119-24. doi: 10.14712/fb2011057030119. PMID 21888835
- [Background] Sekiya I, Muneta T, Horie M, Koga H. Arthroscopic Transplantation of Synovial Stem Cells Improves Clinical Outcomes in Knees With Cartilage Defects. Clin Orthop Relat Res. 2015 Jul;473(7):2316-26. doi: 10.1007/s11999-015-4324-8. Epub 2015 Apr 30. PMID 25925939
- [Background] Zhu H, Jiang XX, Wu Y, Liu YL, Li XS, Zhang Y, Mao N. [Identification of mesenchymal stem cells derived from rheumatoid arthritis synovial fluid and their regulatory effect on osteoblast formation]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2009 Aug;17(4):977-80. Chinese. PMID 19698242
- [Background] Sekiya I, Ojima M, Suzuki S, Yamaga M, Horie M, Koga H, Tsuji K, Miyaguchi K, Ogishima S, Tanaka H, Muneta T. Human mesenchymal stem cells in synovial fluid increase in the knee with degenerated cartilage and osteoarthritis. J Orthop Res. 2012 Jun;30(6):943-9. doi: 10.1002/jor.22029. Epub 2011 Dec 6. PMID 22147634
- [Background] Matsumoto T, Kubo S, Sasaki K, Kawakami Y, Oka S, Sasaki H, Takayama K, Tei K, Matsushita T, Mifune Y, Kurosaka M, Kuroda R. Acceleration of tendon-bone healing of anterior cruciate ligament graft using autologous ruptured tissue. Am J Sports Med. 2012 Jun;40(6):1296-302. doi: 10.1177/0363546512439026. Epub 2012 Mar 16. PMID 22427618
- [Background] Radice F, Yanez R, Gutierrez V, Rosales J, Pinedo M, Coda S. Comparison of magnetic resonance imaging findings in anterior cruciate ligament grafts with and without autologous platelet-derived growth factors. Arthroscopy. 2010 Jan;26(1):50-7. doi: 10.1016/j.arthro.2009.06.030. PMID 20117627
- [Background] Berdis AS, Veale K, Fleissner PR Jr. Outcomes of Anterior Cruciate Ligament Reconstruction Using Biologic Augmentation in Patients 21 Years of Age and Younger. Arthroscopy. 2019 Nov;35(11):3107-3113. doi: 10.1016/j.arthro.2019.05.047. Epub 2019 Aug 19. PMID 31439458
- [Background] Looney AM, Leider JD, Horn AR, Bodendorfer BM. Bioaugmentation in the surgical treatment of anterior cruciate ligament injuries: A review of current concepts and emerging techniques. SAGE Open Med. 2020 May 12;8:2050312120921057. doi: 10.1177/2050312120921057. eCollection 2020. PMID 32435488
- [Background] Wang C, Hu Y, Zhang S, Ruan D, Huang Z, He P, Cai H, Heng BC, Chen X, Shen W. Application of Stem Cell Therapy for ACL Graft Regeneration. Stem Cells Int. 2021 Aug 2;2021:6641818. doi: 10.1155/2021/6641818. eCollection 2021. PMID 34381504
- [Background] Kim K, Zhao R, Doi A, Ng K, Unternaehrer J, Cahan P, Huo H, Loh YH, Aryee MJ, Lensch MW, Li H, Collins JJ, Feinberg AP, Daley GQ. Donor cell type can influence the epigenome and differentiation potential of human induced pluripotent stem cells. Nat Biotechnol. 2011 Nov 27;29(12):1117-9. doi: 10.1038/nbt.2052. PMID 22119740
- [Background] Musial-Wysocka A, Kot M, Majka M. The Pros and Cons of Mesenchymal Stem Cell-Based Therapies. Cell Transplant. 2019 Jul;28(7):801-812. doi: 10.1177/0963689719837897. Epub 2019 Apr 24. PMID 31018669
- [Background] Takeuchi H, Niki Y, Matsunari H, Umeyama K, Nagashima H, Enomoto H, Toyama Y, Matsumoto M, Nakamura M. Temporal Changes in Cellular Repopulation and Collagen Fibril Remodeling and Regeneration After Allograft Anterior Cruciate Ligament Reconstruction: An Experimental Study Using Kusabira-Orange Transgenic Pigs. Am J Sports Med. 2016 Sep;44(9):2375-83. doi: 10.1177/0363546516650881. Epub 2016 Jun 21. PMID 27329998
- [Background] Davies GJ, McCarty E, Provencher M, Manske RC. ACL Return to Sport Guidelines and Criteria. Curr Rev Musculoskelet Med. 2017 Sep;10(3):307-314. doi: 10.1007/s12178-017-9420-9. PMID 28702921
- [Background] Grassi A, Bailey JR, Signorelli C, Carbone G, Tchonang Wakam A, Lucidi GA, Zaffagnini S. Magnetic resonance imaging after anterior cruciate ligament reconstruction: A practical guide. World J Orthop. 2016 Oct 18;7(10):638-649. doi: 10.5312/wjo.v7.i10.638. eCollection 2016 Oct 18. PMID 27795945
- [Background] Lundberg M, Styf J, Jansson B. On what patients does the Tampa Scale for Kinesiophobia fit? Physiother Theory Pract. 2009 Oct;25(7):495-506. doi: 10.3109/09593980802662160. PMID 19925172
- [Background] Brodke DJ, Saltzman CL, Brodke DS. PROMIS for Orthopaedic Outcomes Measurement. J Am Acad Orthop Surg. 2016 Nov;24(11):744-749. doi: 10.5435/JAAOS-D-15-00404. PMID 27661391
- [Background] O'Connor CM, Ring D. Correlation of Single Assessment Numeric Evaluation (SANE) with other Patient Reported Outcome Measures (PROMs). Arch Bone Jt Surg. 2019 Jul;7(4):303-306. PMID 31448305
- [Background] Parekkadan B, Milwid JM. Mesenchymal stem cells as therapeutics. Annu Rev Biomed Eng. 2010 Aug 15;12:87-117. doi: 10.1146/annurev-bioeng-070909-105309. PMID 20415588
- [Background] Yoshihara M, Hayashizaki Y, Murakawa Y. Genomic Instability of iPSCs: Challenges Towards Their Clinical Applications. Stem Cell Rev Rep. 2017 Feb;13(1):7-16. doi: 10.1007/s12015-016-9680-6. PMID 27592701
- [Background] Takayama K, Kawakami Y, Mifune Y, Matsumoto T, Tang Y, Cummins JH, Greco N, Kuroda R, Kurosaka M, Wang B, Fu FH, Huard J. The effect of blocking angiogenesis on anterior cruciate ligament healing following stem cell transplantation. Biomaterials. 2015 Aug;60:9-19. doi: 10.1016/j.biomaterials.2015.03.036. Epub 2015 May 14. PMID 25965282

DOCUMENTS (2):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT05582226/Prot_000.pdf
  • Informed Consent Form (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT05582226/ICF_001.pdf